CLINICAL TRIAL: NCT05427266
Title: Laparoscopic Transversus Abdominis Plane Block (LTAP) (Tap Block) for Appendicectomy Versus Standard Port Site Treatment
Brief Title: Laparoscopic Transversus Abdominis Plane Block (LTAP) for Appendicectomy Versus Standard Port Site Treatment
Acronym: TapBlock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/31
Record Dates: First submitted 2022-06-09; First posted 2022-06-22 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Pain; Appendicitis; Surgery; Analgesia; Laparoscopic; Bupivacaine
MeSH Terms: conditions — Pain; Appendicitis; Agnosia

STUDY DESIGN:
Intervention Model Description: Multi centre Single blinded randomised control trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinded randomised control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group - Tap Block (Other): Study Group: Study group: Laparoscopic Transversus Abdominis Plane in four points: above and below the umbilicus in both right and left sides; dose calculation 2.5mg per body weight.
  After the appendicectomy is done and just before withdrawing port and deflating the abdomen, the operating surgeon will advance a needle into the abdominal wall to the level of the preperitoneal space. Once the needle tip is seen, it is withdrawn slowly and gently about 0.5cm above/superficial to the transversus abdominis (TA) muscle. The surgeon then infiltrates the local anaesthetic into the plane, and the right plane is confirmed by visualising a uniform protrusion downwards of the TA muscle fibres (Doyle's bulge). Seeing a preperitoneal or muscle blister laparoscopically indicates that the infiltration is deeper to this plane, and the needle should be withdrawn more superficially.
  Interventions: Other: Tap Block - Bupivacaine
- Control Group - Standard port site infiltration (Other): Patients will be randomised after diagnosis either clinically or radiologically of appendicitis (both complicated and uncomplicated) Control Group _ standard port site infiltration using 0.25% plain bupivacaine. The dose is calculated to 2.5mg/per kg body weight. After the appendicectomy is done, after removal of ports and deflating the abdomen, the total calculated dose volume will be infiltrated into the subcutaneous plane at the umbilicus and the other 2 ports sites
  Interventions: Other: Tap Block - Bupivacaine

INTERVENTIONS:
Other: Tap Block - Bupivacaine — The medicinal product for both groups is the same - Bupivacaine. The mode of administration is what this study is reviewing: Control group (Standard port site infiltration) and Study Group - Laparoscopic Transversus Abdominis Plane Block (LTap Block)

SUMMARY:
This study aims to compare Laparoscopic assisted LTAP (Transversus Abdominis Plane) to standard port-site infiltration in terms of post-operative visual analogue scores (VAS) for pain at 3, 6, 12 and 24 hours following laparoscopic appendicectomy Tap Block is a standard conventional analgesia protocol for laparoscopic appendicitis used in Beaumont Hospital, and other hospitals throughout Ireland.

The medicinal product for both groups is the same - Bupivacaine. The mode of administration is what this study is reviewing: Control group (Standard port site infiltration) and Study Group - Laparoscopic Transversus Abdominis Plane Block

DETAILED DESCRIPTION:
Title: Randomised Controlled Trial to compare Laparoscopic Transversus Abdominis Plane Block (LTAP) for appendicectomy versus standard treatment Short title: (TAP Block Study) Laparoscopic Transversus Abdominis Plane Block for Appendicectomy - Single-Blinded Randomised controlled study

Objectives: Primary objectives:

To compare LTAP to standard port-site infiltration in terms of post-operative visual analogue scores (VAS) for pain at 3,6, 12 and 24 hours following laparoscopic appendicectomy

Secondary objectives:

Post-operative Opioid requirement Time to first mobilisation post-operatively Length of stay in hospital Quality of Life Questionnaire (at 1 week and 1 month post discharge) (EQ5DL)

Type of trial: Multi centre Single blinded randomised control trial. (Beaumont Hospital and 3 other Dublin Hospitals) Trial design and methods: Study design: randomised controlled Single blind study. Patients will be allocated to one of two parallel groups in a 1:1 fashion. Patients and data analysts will be blinded as to modalities and group allocations. Surgeons and anaesthetists will be made aware of group allocations post randomisation.

Study groups and techniques of anaesthesia:

Control Group: standard port site infiltration using 0.25% plain bupivacaine. The dose is calculated to 2.5mg/kg per body weight. After the appendicectomy is done, after removal of ports and deflating the abdomen, the total calculated dose volume will be infiltrated into the subcutaneous plane at the umbilicus and the other 2 ports sites .

Study group: LTAP block in four points: above and below the umbilicus in both right and left sides; dose calculation 2.5mg per body weight.

After the appendicectomy is done and just before withdrawing port and deflating the abdomen, the operating surgeon will advance a needle into the abdominal wall to the level of the preperitoneal space. Once the needle tip is seen, it is withdrawn slowly and gently about 0.5cm above/superficial to the transversus abdominis (TA) muscle. The surgeon then infiltrates the local anaesthetic into the plane, and the right plane is confirmed by visualising a uniform protrusion downwards of the TA muscle fibres (Doyle's bulge). Seeing a preperitoneal or muscle blister laparoscopically indicates that the infiltration is deeper to this plane, and the needle should be withdrawn more superficially.

Trial duration per participant: 1 month (follow up calls 1 week and 1 month post discharge) Estimated total trial duration: It is estimated that the trial recruitment will take 1 year (based on appendicitis admission rates in both Beaumont Hospital and 3 other Dublin Hospitals). The trial will end once the final patient's follow-up is completed and assessed.

Planned trial sites: Multi-site - sites Beaumont Hospital and 3 other Dublin hospitals Total number of participants planned: 172 86 Control Group 86 Study Group - TAP Block

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for follow up telephone follow up
* Male or female, aged over 18
* Diagnosed either clinically or radiologically (CT/US/MRI) with appendicitis
* Uncomplicated or complicated appendicitis
* Undergoing laparoscopic appendicitis surgery only
* Must be fluent in English in order to complete telephone follow up questionnaire
* Fulfillment of each criteria must be clearly evidenced (in lab reports or correspondence) and/or documented in the medical records.

Exclusion Criteria:

* Male or female under the age or 18
* Laparoscopic converted to open appendicectomy (during surgical procedure)
* Open appendicectomy (planned)
* Pregnancy.
* Females must not be breastfeeding
* Known allergic reactions to components of the study product(s) )
* Not fluent in English - which would prevent participants to complete follow up telephone questionnaire
* Malignant appendicitis
* Spinal Anaesthesia, Epidural analgesia catheter or injections, Post-operative requirements for patient controlled analgesia (PCA)
* Right hemicolectomy or any concomitant or simultaneous intervention
* Allergy or hypersensitivity to any of the components of Bupivacaine
* Presence of any other illness or condition that renders the patient unsuitable for trial participation in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assessing pain post laparoscopic appendicectomy using Visual analogue score (VAS score) | Assessing change in pain score post extubation at 3 hours, 6 hours, 12 hours and 24 hours.
  Assessing any change in pain score from a scale of 1 to 10 (1 being the worst pain and 10 no pain) using VAS score template

SECONDARY OUTCOMES:
Post-operative Opioid requirement | Assess opioid requirement post operatively in the first 24 hours
  Review of opioid requirement (dosage and time delivered) post operatively in both arms to assess if there is a difference in requirement
Time to first mobilisation post-operatively | Assess time to mobility in the first 24 hours post operatively
  Assess any difference in time to mobilization post operatively in both arms
Length of stay in hospital | Assess length of stay from admission to discharge
  Assess if there are any difference in hospital stay in both arms
Quality of Life Questionnaire (at 1 week and 1 month post discharge) (EQ5DL) | 1 week (up to 7 days) and 1 month up to 30 days post discharge from hospital
  Phone follow up with EQ5DL questionnaire by research nurse to assess quality of life and overall satisfaction in both arms. The EQ-5DL The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Hill, Principal Investigator — Royal College of Surgeons in Ireland

IPD SHARING:
Plan to Share IPD: Yes
Paper will be published in surgical journals
Time Frame: 6 months after close of study when analyses is completed
Access Criteria: All findings will be published in surgical journals

REFERENCES:
- [Derived] Daly GR, Dowling GP, Hembrecht S, O'Grady S, Hegarty A, Roche T, Orsi G, Pierre A, Calpin GG, Neary C, Hehir CM, Hill GJ, O'Brien A, Duggan WP, Davey MG, Stephens IJB, Kennedy ND, Brennan O, Hayes C, Al Azzawi M, Balasubramanian I, McGuire A, Zaborowski AM, Reynolds IS, Loughlin P, Allen M, Power C, Butt A, Boland MR, McCawley N, Burke JP, Robb WB, Mastrosimone A, Arumugasamy M, Prins H, Beddy D, Kerin MJ, McNamara DA, Kearney D, Sorensen J, Curley GF, Abd El Wahab S, Hill ADK. Laparoscopic-assisted transversus abdominis plane block versus port-site infiltration in appendicectomy: multicentre randomized clinical trial. Br J Surg. 2025 Dec 24;113(1):znaf257. doi: 10.1093/bjs/znaf257. PMID 41511871